CLINICAL TRIAL: NCT00001006
Title: A Phase One Study of AS-101 in Patients With Acquired Immune Deficiency Syndrome (AIDS) or AIDS-Related Complex (ARC)
Brief Title: A Study of AS-101 in Patients With AIDS or AIDS Related Complex (ARC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 046; 11020 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Infusions, Intravenous; Immunologic Surveillance; Drug Evaluation; Adjuvants, Immunologic; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; ammonium trichloro(dioxoethylene-O,O'-)tellurute
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — ammonium trichloro(dioxoethylene-O,O'-)tellurate

INTERVENTIONS:
Drug: AS-101

SUMMARY:
To determine the toxic effects of AS-101 at various doses in patients with AIDS or AIDS related complex. Also to determine the effect of various doses of AS-101 on immune functions and the occurrence of infections in these patients. AIDS is a viral disease that is characterized by a loss of some immune function and the development of frequent, eventually fatal, infectious diseases. Although zidovudine (AZT) has prolonged survival in some patients with AIDS, AZT is quite toxic and there is a need for more effective and less toxic drugs. AS-101 is a synthetic organic compound containing the metal tellurium that is being tested because in laboratory studies it improved immune functions.

DETAILED DESCRIPTION:
AIDS is a viral disease that is characterized by a loss of some immune function and the development of frequent, eventually fatal, infectious diseases. Although zidovudine (AZT) has prolonged survival in some patients with AIDS, AZT is quite toxic and there is a need for more effective and less toxic drugs. AS-101 is a synthetic organic compound containing the metal tellurium that is being tested because in laboratory studies it improved immune functions.

Patients are given intravenous infusions of AS-101 3 times a week for 12 weeks. The first group of 6 patients receives a dose that did not cause toxic effects in a preliminary study. If no adverse effects occur, the next 6 patients receive a higher dose level and so on, until an optimum dose has been reached. The investigators will determine the optimum dose based on the type and severity of adverse effects experienced by the patients on the study and by the effect of the drug on the immune function of the patient and its effect on the HIV infection. Samples of blood and urine are taken periodically during the study and skin tests are performed 3 times to aid in the evaluation of AS-101. Patients receive standard treatment for any infections that develop during the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Inhaled pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Ketoconazole.
* Standard outpatient therapy for infections developing during the trial.
* Oral acyclovir for up to 7 days.

Patients must have:

* Antibody to HIV by ELISA.
* AIDS or AIDS related complex (ARC).
* T4 cell count < 400 cells/mm3 on 2 determinations at least 72 hours apart.

Prior Medication:

Allowed:

* Inhaled pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Ketoconazole.
* Oral acyclovir for up to 7 days.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active opportunistic infection or malignancy requiring concurrent treatment.
* Serious medical problems, such as diabetes, renal disease, ASHD, or hypertension, which would complicate interpretation of treatment results.
* Transfusion requirements exceeding 2 transfusions per month in order to achieve hemoglobin > 9 g/dl.

Concurrent Medication:

Excluded:

* Treatment for active opportunistic infection or malignancy.
* Systemic antiviral preparations.
* Immunosuppressive agents.
* Immunostimulation therapy.
* Specific therapy for Kaposi's sarcoma or other malignancies.

Concurrent Treatment:

Excluded:

* More than 2 units of red blood cell transfusions per month in order to achieve hemoglobin > 8 g/dl.

Patients unlikely or unable, for reasons such as distance from the hospital or psychological considerations, to comply with the requirements of the protocol, especially in regard to regular attendance for treatment, are excluded.

Prior Medication:

Excluded:

* Systemic antiviral preparations.
* Isoprinosine.
* Excluded with 1 month of study entry:
* Immunosuppressive agents.
* Immunomodulators.

Prior Treatment:

Excluded:

* Immunostimulation therapy, such as BCG vaccine.

Active drug or alcohol abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Study Completion 1993-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sacks HS, Study Chair; Hassett J, Study Chair
Locations (1):
- Mount Sinai Med Ctr, New York, New York, United States

REFERENCES:
- [Background] Lewi DS, Acceturi CA, Diaz RS, Lofty C, Sader H. AS 101: tolerability, safety and clinical efficacy in HIV positive patients with advanced disease. Int Conf AIDS. 1992 Jul 19-24;8(3):100 (abstract no PuB 7310)